CLINICAL TRIAL: NCT01208350
Title: Testing Strategies to Encourage Weight Loss in an Employer Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other); incentaHEALTH (Industry); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 812193; RC2AG036592 (NIH)
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2012-09

CONDITIONS: Weight Loss
Keywords: Weight Loss; Motivation; Workplace; Web platform
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Individual payout
- 2 (Experimental)
  Interventions: Behavioral: Group-based payout
- 3 (Active Comparator)
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: No intervention — Monthly weigh-ins for 6 months without financial incentives associated with weight loss, and follow-up weigh-in at 9 months
  Arms: 3
Behavioral: Group-based payout — Monthly weigh-ins for 6 months where five sequential participants, randomized to this condition, will be joined into virtual groups where individual rewards for weight loss are dependent on the weight loss of others in the group, with follow-up weigh in at 9 months
  Arms: 2
Behavioral: Individual payout — Monthly weigh-ins for 6 months and if monthly goals are met, participants receive payout at the end of the month, with follow-up weigh-in at 9 months
  Arms: 1

SUMMARY:
This is a 3-arm pilot randomized controlled trial to evaluate the effectiveness of two novel ways of structuring financial incentives to motivate and sustain long-term weight loss. The study will recruit eligible employees at Children's Hospital of Philadelphia (CHOP) to participate in a 6-month weight loss program and an additional 3-month follow-up period. The primary outcome measure in this randomized control trial will be pounds of weight lost between baseline and 6 months. The goal of this study is to evaluate whether a novel financial incentive program delivered through a workplace can effectively encourage sustained weight loss among obese employees.

The study hypotheses are 1) mean weight loss will be greater in all the intervention groups compared to the control group by the end of the 24-week intervention period; and 2) individuals in the intervention groups will have a lower mean weight at the end of the 12-week follow-up period than individuals in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 (inclusive)
* BMI between 30 and 40 (inclusive)

Exclusion Criteria:

* Inability to consent
* Illiteracy and/or inability to speak, read, and write English
* Participation in another research study
* Current treatment for drug or alcohol use
* Consumption of ≥ 5 alcoholic drinks per day
* Myocardial infarction or stroke within the past 6 months
* Current addiction to prescription medicines or street drugs
* Serious psychiatric diagnoses (e.g., severe major depressive disorder, bipolar disorder, schizophrenia)
* Pregnant or currently breastfeeding
* Diabetic and using any medicine besides metformin to control blood glucose
* Metastatic cancer
* Unstable medical conditions that would likely prevent the subject from completing the study
* Previous diagnosis of an eating disorder
* History of unsafe weight loss behaviors such as binging or the use of laxatives

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in weight between baseline and six months | 24 weeks

SECONDARY OUTCOMES:
usability of a newly developed web portal and its feasibility for future randomized clinical trials aimed at changing health-related behaviors | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Study Chair — University of Pennsylvania; Jeffrey T Kullgren, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kullgren JT, Troxel AB, Loewenstein G, Asch DA, Norton LA, Wesby L, Tao Y, Zhu J, Volpp KG. Individual- versus group-based financial incentives for weight loss: a randomized, controlled trial. Ann Intern Med. 2013 Apr 2;158(7):505-14. doi: 10.7326/0003-4819-158-7-201304020-00002. PMID 23546562